CLINICAL TRIAL: NCT05578040
Title: Survey on the Changing Temperature of the Skin Surface in the Neck Area When Auricular Acupressure at Cervical Vertebra Acupoints in Healthy Volunteers: a Randomized Controlled Trial
Brief Title: Skin Surface's Temperature Changes When Auricular Acupressure at Cervical Vertebra Acupoints in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bui Pham Minh Man (Other)
Responsible Party: Sponsor-Investigator, Bui Pham Minh Man, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 676/HDDD-DHYD
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Auricular Acupressure

STUDY DESIGN:
Intervention Model Description: A randomized controlled and single blinded trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Left AH13 acupoint (left cervical vertebra) (Experimental): Participants received sham auricular acupressure by adhesive patches without Vaccaria seed at the left auricular cervical vertebra acupoint and auricular acupressure Vaccaria seed at the left auricular cervical vertebra acupoint after 1 week. At each time, the skin surface temperature of the neck area will be recorded.
  Interventions: Procedure: Auricular acupressure
- Group B: RIght AH13 acupoint (right cervical vertebra) (Experimental): Participants received sham auricular acupressure by adhesive patches without Vaccaria seed at the right auricular cervical vertebra acupoint - and auricular acupressure Vaccaria seed at the right auricular cervical vertebra acupoint after 1 week. At each time, the skin surface temperature in the neck area will be recorded.
  Interventions: Procedure: Auricular acupressure

INTERVENTIONS:
Procedure: Auricular acupressure — To conduct this intervention, we used adhesive patches without Vaccaria seed to sham auricular acupressure at the cervical vertebra acupoint in the first trial phase and auricular acupressure at the cervical vertebra acupoint in the other two trial phases in 2 groups of auricular acupressure acupoints of the left and right cervical vertebra.

SUMMARY:
Auricular acupressure is one of the acupuncture techniques on the ear, which is a method of impacting on acupoints with force and without using needles to help diagnose and treat physical and psychosomatic dysfunctions. Some studies prove that the acupoints on the pinna have a corresponding relationship with the areas of the body, and when acting on the acupoints can change the temperature of the corresponding area. Chronic neck pain is closely related to the decline in subcutaneous microcirculation, where heat transfer from deep within the body to the surface of the skin is carried out by the dermal vascular system. When blood flow through the venous network is high, heat is carried from the deep to the skin and vice versa. Therefore, to understand the role of cervical vertebra acupoints in neck pain, the study wants to demonstrate the correlation when auricular acupressure at cervical vertebra acupoints and the skin surface temperature of the neck area.

DETAILED DESCRIPTION:
Participants and Methods: A randomized controlled trial is conducted by surveying the change in temperature in the neck area respectively when auricular acupressure is applied to the left and right cervical vertebra acupoints compared with the sham auricular acupressure group in each side of the ear in healthy volunteers. A total of 60 participants were randomly assigned to 2 groups (A and B) and the allocation was 1:1. In group A: participants received sham auricular acupressure at the left AH13 acupoint (left cervical vertebra) of the ear and auricular acupressure after 1 week. In group B: participants received sham auricular acupressure at the right AH13 acupoint (right cervical vertebra) of the ear and auricular acupressure after 1 week. The primary outcome was change in temperature in the neck area respectively when auricular acupressure is applied to the left and right cervical vertebra acupoints compared with the sham auricular acupressure group. This trial will be performed as randomized, controlled, and single blinded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, regardless of gender or profession
* Age between enough 18 and 30 years old.
* No psychological problems (anxiety, depression, stress): assessed according to DASS 21 score, with stress score < 15 points.
* Vital signs within normal limits:

  * Heart rates from 60 to 100 beats/minute
  * Systolic blood pressure between 90 and 139 mmHg
  * Diastolic blood pressure between 60 and 89 mmHg
  * Body temperature: 36.59 ± 0.43 0C
  * Breathing rate: 16 ± 3 times/minute
* Voluntarily agree to participate in the research and sign the consent form to participate in the research after being advised by the researcher and clearly explaining the rights and obligations when participating in the research.
* Not currently participating in other intervention studies.
* No knowledge and experience of auricular acupressure method.

Exclusion Criteria:

* Having an inflammatory injury in the site of the skin to be investigated.
* Using heat therapy, for example, massage, cupping therapy, and acupuncture in the site of the skin to be investigated within 24h.
* Applying chemical or pharmaceutical products to the site of the skin to be surveyed before conducting the study.
* Other diseases that could affect or interfere with outcomes, including the common cold or flu.
* Having neck pain, dermatitis, skin infection, and wound in the survey area.
* Having diseases that change the body temperature, like hyperthyroidism, and hypothyroidism.
* Taking stimulants (alcohol, beer, coffee, tobacco) within 24h.
* Staying up at night or having insomnia before the day of the study.
* Playing sport within 2h.
* Pregnant woman or woman in the period.
* Are taking some sleeping pills, sedatives, or drugs that cause vasodilation, lower blood pressure
* Anxiety, depression, and stress before conducting the study with DASS 21 score > 15 points.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Survey the change in temperature in the neck area respectively when auricular acupressure is applied to the left and right cervical vertebra acupoints compared with the sham auricular acupressure group | During procedure
Change the temperature of skin surface in the neck area when using auricular acupressure at cervical vertebra acupoints on each side of the ear | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- See also: Guan L, Li G, Yang Y, Deng X, Cai PJNRR. Infrared thermography and meridian-effect evidence and explanation in Bell's palsy patients treated by moxibustion at the Hegu (LI4) acupoint: Overall regulation or a specific target?. 2012;7(9):680. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4347008/
- See also: Song X, Zhang DJZZjCA, Moxibustion. Study on the manifestation of facial infrared thermography induced by acupuncturing Guangming (GB 37) and Hegu (LI 4). 2010;30(1):51-54 — https://www.scirp.org/%28S%28lz5mqp453edsnp55rrgjct55%29%29/reference/referencespapers.aspx?referenceid=2755362